### INFORMATION SHEET FOR INVOLVEMENT FOCUSS FEEDBACK INTERVIEW

#### YALE UNIVERSITY

Project Title: Feedback and Outcomes for Clinically Useful Student Services (FOCUSS)

# Principal Investigator (the person who is responsible for this project):

Elizabeth H. Connors 389 Whitney Ave, New Haven, CT 06511

### **FOCUSS Project Summary:**

- You are involved in the FOCUSS project because you provide school-based mental health treatment services and your district administrators have consented to district-wide participation.
- The purpose of FOCUSS is to increase clinicians' use of student and parent-reported measures in school mental health. This practice is called "measurement-based care" or "MBC."
- FOCUSS project activities this year have included:
  - A 3-hour interactive training on measurement-based care in schools.
  - Six, 60-minute, monthly post-training consultation calls for six months following the training.
  - Four, 30-minute online feedback surveys from clinicians.
  - Collecting student progress data using Better Outcomes Now (BON) with at least five (5) of your students.
  - Parent recruitment. We will ask you to refer at least five (5) parents to the research study component of this project.

### Feedback Interview Summary (new activity):

- Because you are involved in the FOCUSS project, you have been randomly selected to participate in a 20-30 minute feedback interview.
- The interview will take place via Zoom, and will be recorded.
- Interviews have been added to the FOCUSS project activities to help us gather more in-depth feedback on the clinician's experience this year, to add to what we learned in the online feedback surveys.
- Interview questions include your experiences about obstacles and supports related to measurement-based care, parent engagement, and recommendations for FOCUSS next year.
- We do not expect any risks from taking part in this project.
- You may benefit from taking part in this interview by sharing your experiences and recommendations to improve project improvements for yourself and other clinicians in future years.
- If you are interested in learning more about the interviews, please continue reading, or have someone read to you, the rest of this document. Ask study staff questions about anything.

### Are there any costs to involvement? Will I be paid for involvement?

There is no cost to your involvement in this study. You will receive a \$25 Amazon gift card two to three weeks after completion.

## How will you keep my data safe and private?

Your participation in an interview and your repsonses responses will be kept confidential and will not impact your employment or performance review in any way. Only the researchers involved in this study and those responsible for research oversight (such as representatives of the Yale University Human Research Protection Program, the Yale University Institutional Review Boards, and others) will have

access to any information that could identify you that you provide. We will share it with others if you agree to it or when we have to because U.S. or State law requires it. For example, we will tell somebody if we learn that you are hurting a child or an older person.

Your district leadership will not know whether or not you decide to participate.

Your interview responses will be added to that of other clinicians, summarized and shared in a deidentified manner with your district leadership for the purposes of improving FOCUSS next year. We will send you the summary for your reference, feedback and to ensure accuracy before it is provided to your district leadership.

When we publish the results of the research or talk about it in conferences, we will not use your name. If we want to use your name, we will ask you for your permission. We will also share information about you with other researchers for future research, but we will not use your name or other identifiers. We will not ask you for any additional permission.

# Who should I contact if I have questions?

Please feel free to ask about anything you don't understand.

If you have questions later or if you have a research-related problem, you can call the Principal Investigator, Dr. Elizabeth Connors, at 203-789-7645 x116 or the PI's research assistant, Sophia Selino, at 203-789-7645 x184.

If you have questions about your rights as a research participant, or you have complaints about this research, you call the Yale Institutional Review Boards at (203) 785-4688 or email <a href="mailto:hrpp@yale.edu">hrpp@yale.edu</a>.